CLINICAL TRIAL: NCT03474419
Title: Evaluation of the Satisfaction of the Patients Operated for a Mild Hyperplasie of the Prostate by Laser in Ambulatory Surgery
Status: Withdrawn | Type: Observational
Why Stopped: The principal investigator decide to stop the sudy.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PROSTATAMBU
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Laser Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laser surgery — laser surgery

SUMMARY:
Every year more than 70 000 interventions for prostatic adenoma are realized. Several type of surgery are realized going of the ambulatory to longer hospital lengths of stay. There are also several techniques.However it appears that ambulatory surgery is less costly. The arguments of surgeons are patients reluctance or the difficulty to manage in case of complication.

The aim of the study is to show that there is a good acceptance from patient with a good level of satisfaction at day 30.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18
* patient with benign prostatic hyperplasia
* ambulatory eligibility

Exclusion Criteria:

* recused for ambulatory surgery
* Patients operated by surgeons not having ended their learning curve.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only male
Study Population: 33 patients selected in the 6 center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | Day 30
  analogic scale (0 to 10)